CLINICAL TRIAL: NCT04477083
Title: Development and Validation of "Ready-to-Use" Inhalable Forms of Hydroxychloroquine for Treatment of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ibrahim M. El-Sherbiny, PHD, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: inhalable HCQ
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Hydroxychloroquine Adverse Reaction
Keywords: Covid19; Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: The first 20 consecutive patients (group A) will be treated by oral antibiotics, supportive treatment and inhalable hydroxychloroquine (HCQ). (In day 1, an inhaled hydroxychloroquine sulfate dose of 12 mg will be taken via nebulization three times/day (TID) as a loading dose. Then, starting from day 2, same dose of 12 mg of inhaled hydroxychloroquine will be taken twice/day (BID) as maintenance dose for 5 days. The subsequent 20 consecutive patients (group B) will receive the same treatment of group A but without inhalable hydroxychloroquine (HCQ). At day 7, all patients of both groups will be evaluated by clinical, laboratory and chest CT parameters. Patients of group B who still show no clinical, laboratory or radiological improvement will continue treatment by adding inhalable hydroxychloroquine (HCQ). for another 7 days and re-evaluated at day 14. Patients of group A who still show no significant improvement at day 7 only will be re-checked at day 14.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhalable hydroxychloroquine (HCQ). (Active Comparator): supportive and symptomatic treatment and inhalable hydroxychloroquine (HCQ).
  Interventions: Drug: inhalable hydroxychloroquine (HCQ)
- Placebo (Placebo Comparator): supportive and symptomatic treatment
  Interventions: Drug: supportive and symptomatic treatment

INTERVENTIONS:
Drug: inhalable hydroxychloroquine (HCQ) — inhalable hydroxychloroquine (HCQ) plus supportive and symptomatic treatment
  Arms: inhalable hydroxychloroquine (HCQ).
Drug: supportive and symptomatic treatment — supportive and symptomatic treatment
  Arms: Placebo

SUMMARY:
In this project, we aimed at developing new "Ready-to-Use" inhalable forms of HCQ that can be used directly through nebulization or using dry powder inhalers (DPIs). These inhaled forms would allow a simple and direct delivery of the drug (HCQ) specifically towards the throat and the lung which are the main sites for the COVID-19 viral infection. Hence, the drug can be available at higher concentrations in the throat and lungs as compared with the currently used treatment protocols, while minimizing the drug systemic concentrations and its presence in other body organs, and thus enhancing the drug efficacy with significantly limiting its side effects. Besides, using inhalable forms can be more convenient to patients suffering from gastrointestinal complications from the disease that can limit the absorption of oral forms. Moreover, the proposed inhalable forms are designed in such a way to hide the drug from the immune system (confer stealth characteristics) using FDA-approved excipients to minimize/avoid any immune response towards the drug as was noted towards it in its oral form that's used in the treatment protocol of COVID-19. In addition, the inhaled formulations will be designed to maintain the overall simplicity and scalability of the preparation which is critical during this urgent pandemic situation. The cost of the final formulation is also taken into consideration since the drug is intended for treatment of thousands or probably millions of patients around the world including countries with limited economic capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Laboratory (RT-PCR) positive of SARS-COV-2 (Moderate cases)
* Chest CT with pneumonia.
* SaO2/SPO2 ratio > 93% or PaO2/FIO2 ratio > 300 mmHg under the condition in the hospital room.
* Welling to participate and able to give fully informed consent

Exclusion Criteria:

* Severe and critical illness.
* Retinopathy and other retinal diseases.
* Arrhythmias.
* QT ≥ 400 msec
* Receiving cardiac drugs
* Severe liver disease.
* Pregnancy or lactation.
* Previous treatment of COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery defined as 3 days afebrile with improved cough and other clinical signs | 15 days
  Time is measured in hours
Time to achieve viral clearance state determined by two successive negative PCR results for two oropharyngeal swabs separated by 48 hours. | 15 days
  Time is measured in hours

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 15 days
  measuring and monitoring the complication between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Outside U.S./Canada, Egypt